CLINICAL TRIAL: NCT01337388
Title: An Observational Study of the Efficacy of RoActemra in Smoking vs Non-smoking Patients With Rheumatoid Arthritis.
Brief Title: An Observational Study of RoActemra/Actemra (Tocilizumab) in Smoking Versus Non-Smoking Patients With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25492
Record Dates: First submitted 2011-04-15; First posted 2011-04-18 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will assess the efficacy and safety of RoActemra/Actemra (Tocilizumab) in smoking versus non-smoking patients with rheumatoid arthritis. Data from patients treated in routine clinical practice with intravenous RoActemra/Actemra will be collected for 12 months each.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, > 18 years of age
* Rheumatoid arthritis, defined as fulfilling at least 4 of 7 American College of Rheumatology (ACR) criteria
* Treatment with RoActemra/Actemra

Exclusion Criteria:

* Participation in interventional clinical studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatoid arthritis patients on treatment with RoActemra/Actemra
Sampling Method: Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2010-08; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change in disease activity score (DAS 28) | 12 months
Treatment patterns (frequency/dosage) and demographics of patients treated with RoActemra/Actemra in routine clinical practice | 36 months

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | 36 months
Quality of life: Health assessment questionnaire Disease Index (HAQ-DI), Functional Assessment of Chronic Illness Therapy- Fatigue (FACIT-Fatigue) questionnaire | 12 months
Rate of patients achieving remission (DAS <2.6) | 36 months
Change in blood lipids | 12 months
Clinical response (DAS 28/blood chemistry/QoL) with or without methotrexate | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (28):
- Norway (9):
  - Ålesund
  - Bergen
  - Drammen
  - Gjettum
  - Kristiansand
  - Levanger
  - Lillehammer
  - Skien
  - Trondheim
- Sweden (19):
  - Eskilstuna
  - Falun
  - Farsta
  - Gothenburg
  - Kalmar
  - Karlstad
  - Kristianstad
  - Linköping
  - Luleå
  - Malmo
  - Oskarström
  - Örebro
  - Östersund
  - Simrishamn
  - Skövde
  - Stockholm
  - Uddevalla
  - Uppsala
  - Västerås